CLINICAL TRIAL: NCT01692769
Title: Randomized Controlled Trial of Intravenous Fluid In Severely Injured Paediatric Trauma Patients: Comparison of Normal Saline Versus Ringer's Lactate
Brief Title: Trial Of Normal Saline Versus Ringer's Lactate In Paediatric Trauma Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 102632
Record Dates: First submitted 2012-09-19; First posted 2012-09-25 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Trauma
Keywords: Trauma; Pediatric; Intravenous Fluid; Normal Saline; Ringer's Lactate
MeSH Terms: conditions — Wounds and Injuries | interventions — Saline Solution; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Saline (Active Comparator): Patients will receive intravenous normal saline for all resuscitation and maintenance fluid for a period of 24 hours commencing on presentation to hospital.
  Interventions: Drug: Normal Saline
- Ringer's Lactate (Active Comparator): Patients will receive intravenous Ringer's Lactate for all resuscitation and maintenance fluid for a period of 24 hours commencing on presentation to hospital.
  Interventions: Drug: Ringer's Lactate

INTERVENTIONS:
Drug: Normal Saline — Patients randomized to Normal Saline arm, will receive intravenous normal saline for all resuscitation and maintenance fluid for a period of 24 hours commencing on presentation to hospital.
  Other Names: 0.9% Normal Saline
  Arms: Normal Saline
Drug: Ringer's Lactate — Patients randomized to Ringer's Lactate arm, will receive intravenous Ringer's Lactate for all resuscitation and maintenance fluid for a period of 24 hours commencing on presentation to hospital.
  Other Names: Lactated Ringers
  Arms: Ringer's Lactate

SUMMARY:
Background: Trauma is a major cause of death in children and teenagers. When young patients have suffered major traumatic injuries, they require intravenous (iv) fluids to keep their blood vessels full and ensure blood flow to vital organs. Current fluid guidelines by International Trauma Committees recommend either Normal Saline (NS) or Ringer's Lactate (RL) as the fluid of choice for these patients. Although these solutions share some similarities in their composition, there are also some significant differences in sodium, chloride and lactate concentrations. Despite these differences in fluid composition, there has never been a study comparing these two fluids in paediatric trauma patients to determine which is optimal. In this study, the investigators aim to determine the optimal fluid choice for trauma resuscitation of young patients.

Hypothesis: The investigators hypothesize that severely injured paediatric trauma patients resuscitated with NS will have optimal blood sodium levels compared to patients resuscitated with RL.

Methods: The investigators will study 50 paediatric trauma patients that will be randomized so that half will randomly receive NS and half will receive RL as their only iv fluid for 24 hours. After 24 hours, the investigators will compare in blood the sodium level, the amount of acid, and the concentrations of inflammation molecules in relation to those whom received NS versus RL.

Expected Results and Significance: Maintaining optimal levels of these biochemical markers is imperative in reducing morbidity and mortality in severely injured paediatric patients. If significant differences are present, the investigators will be able to determine which fluid is preferred and expect these data to complement current trauma resuscitation guidelines.

DETAILED DESCRIPTION:
Background:

Trauma is the major killer of children and adolescents. The care of paediatric trauma patients is guided by the Advanced Trauma Life Support (ATLS) guidelines. Fluid resuscitation is a critical aspect of trauma resuscitation to avoid hypoperfusion and metabolic acidosis, and to maintain adequate oxygen delivery to tissues. ATLS recommends the use of either intravenous Normal Saline (NS) or Ringer's Lactate (RL) in trauma fluid resuscitation. There are currently no recommendations or any studies to suggest which of these two fluids are more appropriate for pediatric trauma patients and their ionic compositions do differ. As such, both solutions have potential benefits and potential complications.

There are three primary issues that relate to choice of solution.

1. Sodium concentration and risk of iatrogenic hyponatremia: NS has higher sodium content relative to RL (154 vs. 130 mmol/L, respectively; normal blood levels are 135-145 mmol/L). Maintenance of a normal or slightly elevated sodium level in paediatric trauma patients is often imperative, given that the vast majority of these patients have significant traumatic brain injury. Hyponatremia can worsen cerebral edema and increase intracranial pressure. In a previous study conducted by us at Children's Hospital, LHSC we reported that paediatric trauma patients in our centre received NS. Despite NS used as the resuscitation fluid, pediatric trauma patients all showed a trend towards low-normal levels of sodium in their blood. Given the lower content of sodium in RL, we question whether NS is superior for maintenance of blood sodium.
2. Chloride concentration and risk of iatrogenic hyperchloremic metabolic acidosis: NS contains significantly more chloride than RL to maintain electro-neutrality (154 vs. 109 mmol, respectively; normal blood levels are 98-108 mmol/L). In contrast, the RL solution replaces 28 mmol/L of chloride with equimolar lactate. As the elevated chloride content in NS is postulated to instigate the undesired consequences of driving blood bicarbonate lower and producing a hyperchloremic metabolic acidosis,6, 7 we question whether NS is inferior to RL for maintenance of blood pH.
3. Exacerbation of trauma-induced inflammation: Trauma results in a systemic inflammatory response (Fraser Lab, unpublished results). Exacerbation of the inflammatory state with non-optimal resuscitation practices might worsen overall outcome. Published data on non-trauma patients suggests that NS administration is pro-inflammatory relative to RL,9 but this possibility has not been studied in paediatric patients, or in any trauma patients. The inflammatory cascade can be assessed in blood by measuring the levels of global inflammatory markers [erythrocyte sedimentation rate (ESR) and C-reactive protein (CRP)] and specific pro-inflammatory mediators elevated by multisystem trauma [interleukin-6 (IL-6), interleukin-8 (IL-8), granulocyte colony stimulating factor (G-CSF) and monocyte chemotactic protein-1 (MCP-1)]. Given the higher inflammatory potential that has been associated with NS, we question whether NS is inferior to RL for minimizing inflammatory cascades.

Hypothesis:

We hypothesize that severely injured paediatric trauma patients resuscitated with NS will have optimal blood sodium levels compared to patients resuscitated with RL, but at the expense of hyperchloremic metabolic acidosis and exaggerated inflammation.

Methodology:

This study will be a prospective, single-blinded, RCT of severely injured paediatric trauma patients admitted to the Children's Hospital, London Health Sciences Centre. While the clinical staff treating the patient will be aware of treatment group, the patient, as well as the laboratory technicians determining the serum changes will be blinded to the fluid administered.

Randomization:

Patients will be immediately randomized to either receive NS or RL as their resuscitation and maintenance fluid for the first 24 hours. Randomization, via selection of sealed envelope based on a computer-generated list, will be done by the trauma resuscitation room intravenous access nurse without delay on arrival. Intravenous access and solution administration occurs as a priority within minutes of arrival to the trauma room.

Clinical Data and Blood Analyses:

All patients included in this study will be entered into the LHSC Trauma Database, comprised of over 400 data elements, by a single, trained Trauma Data Analyst. The database regularly undergoes quality monitoring to ensure the data is complete and is of highest quality. Descriptive analyses and epidemiologic profiles on demographic, clinical and injury data will be undertaken, as we have published previously. A baseline trauma blood panel will be drawn upon presentation to our resuscitation room (Time "0"), and then repeated at 24 hours. Blood measurements for analyses will include serum sodium, chloride, bicarbonate, base excess, osmolality, blood gas, ESR and CRP. An extra blood vial will be taken and stored for batch analyses of pro-inflammatory cytokines by multiplex assay (IL- 6, IL-8, G-CSF and MCP-1). Other interventions will be carried out as per standard of care at the discretion of the Trauma most responsible physician. Any medications or any additional fluids the patients receive will be recorded. The total amount of intravenous fluid received in the first 24 hours will be measured for all patients.

Data Analysis:

Descriptive analyses and epidemiologic profiles on demographic, clinical and injury data will be undertaken, as we have published previously.

Treatment groups will be compared using Mann Whitney U test for the outcome measures at 24 hours, as they are continuous. This will include the primary outcome variable (serum sodium) and the secondary outcome variables (serum chloride, bicarbonate, pH and inflammatory markers: ESR, C-RP, IL-6, Il-8, G-CSF, MCP-1).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric trauma patients with Injury Severity Score greater than 12
* Age 1-17 years
* Trauma within 8 hours

Exclusion Criteria:

* Injury Severity Score less than 12
* Pre-existing renal disease
* On medication that affects serum sodium (i.e diuretic therapy)
* Blood transfusion within first 24 hours
* Operation within first 24 hours
* Oral intake of fluid or solids in first 24 hours

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The difference in serum sodium change over 24 hours between patients receiving NS versus RL | 24 hours

SECONDARY OUTCOMES:
The difference in serum pH | 24 hours
The difference serum chloride | 24 hours
The differences in serum bicarbonate | 24 hours
The differences in serum inflammatory biomarker change: Erythrocyte Sedimentation Rate (ESR) | 24 hours
The differences in serum inflammatory biomarker change: C-Reactive Protein | 24 hours
The differences in serum inflammatory biomarker change: InterLeukin-6 | 24 hours
The differences in serum inflammatory biomarker change InterLeukin-8 | 24 hours
The differences in serum inflammatory biomarker change: G-CSF | 24 hours
The differences in serum inflammatory biomarker change: MCP-1 | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gurinder S Sangha, MD, Principal Investigator — London Health Sciences Centre, University of Western Ontario; Douglas D Fraser, MD, PhD, Principal Investigator — London Health Sciences Centre, University of Western Ontario
Locations (1):
- Children's Hospital, London Health Sciences Centre, London, Ontario, Canada